CLINICAL TRIAL: NCT03861949
Title: Effectiveness of Preoxygenation With Positive Airway Pressure in Non-obese Healthy Patient: a Comparison of the Supine and 25° Head up Position
Brief Title: Effectiveness of Preoxygenation With Positive Airway Pressure: a Comparison of the Supine and 25° Head up Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Yogesh Dhakal, Assistant Professor, Department of Anaesthesiology and Critical Care, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IERB/205/014
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Intubation;Difficult
Keywords: apnea; CPAP; Preoxygenation
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional (No Intervention): preoxygenation done with 100% oxygen in supine position
- Positive-pressure (Experimental): preoxygenation done with 5 cmH2O CPAP (continuous positive airway pressure) in supine position with 100% oxygen
  Interventions: Other: 5 cmH2O CPAP
- Head-up (Experimental): preoxygenation done in 25 degree head-up position with 5 cmH2O CPAP with 100% oxygen
  Interventions: Other: 5 cmH2O CPAP; Other: head-up position

INTERVENTIONS:
Other: 5 cmH2O CPAP
  Arms: Head-up; Positive-pressure
Other: head-up position
  Arms: Head-up

SUMMARY:
Several techniques such as positive airway pressure and head-up tilt during preoxygenation have shown to prolong non-hypoxic apnea period compared to conventional technique. However, uniform recommendations have not yet been made. Therefore, in the present study the investigators attempted to find out the effect of combination of 5 cmH2O CPAP and 25° head up position during preoxygenation.

DETAILED DESCRIPTION:
In this study 60 non-obese healthy adult patients were divided into three groups; Group C receiving preoxygenation in conventional technique, Group S receiving preoxygenation with 5 cmH2O CPAP and Group H receiving preoxygenation in 25° head-up position with 5 cmH2O CPAP. After 3 min of preoxygenation, anesthesia was induced and trachea intubated. After confirming the tracheal intubation by direct visualization, all patients were left apneic in supine position with the tracheal tube exposed to atmosphere till the SpO2 dropped to 92%. The primary outcome compared between the groups was the non-hypoxic apnoeic period (time to fall SpO2 to 92%).

ELIGIBILITY:
Inclusion Criteria:

* adult patients of ASA physical status I and II undergoing surgery under general anaesthesia

Exclusion Criteria:

* anticipated difficult mask ventilation/ intubation
* individuals with significant cardiorespiratory or cerebrovascular disease
* pregnant ladies
* patient with history of epilepsy
* body mass index >25 kg/m2
* hemoglobin <8 gm/dL
* patients who were non-ambulant for >24 h, having SpO2 < 97% while breathing in room air
* phobia to facemask.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06-15 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2015-06-15 (Actual)

PRIMARY OUTCOMES:
non-hypoxic apnoeic period (time to fall SpO2 to 92%) | 2 hours
  After 3 min of preoxygenation, anesthesia was induced and trachea intubated. After confirming the tracheal intubation by direct visualization, all patients were left apneic in supine position with the tracheal tube exposed to atmosphere till the SpO2 dropped to 92%.

SECONDARY OUTCOMES:
Comparison of pH at different time points | 2 hours
  Arterial blood gas analysis was done and the pH at the start of preoxygenation, after preoxygenation and at desaturation (SpO2= 92%) were compared.
Comparison of PaO2 at different time points | 2 hours
  Arterial blood gas analysis was done and the PaO2 at the start of preoxygenation, after preoxygenation and at desaturation (SpO2= 92%) were compared.
Comparison of PaCO2 at different time points | 2 hours
  Arterial blood gas analysis was done and the PaCO2 at the start of preoxygenation, after preoxygenation and at desaturation (SpO2= 92%) were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Balkrishna Bhattarai, Professor, Principal Investigator — B.P. Koirala Institute of Health Sciences; Sindhu Khatiwada, Professor, Principal Investigator — B.P. Koirala Institute of Health Sciences; Asish Subedi, Dr, Principal Investigator — B.P. Koirala Institute of Health Sciences

IPD SHARING:
Plan to Share IPD: No